CLINICAL TRIAL: NCT00468546
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Study to Evaluate the Safety and Efficacy of Rituximab in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-TNF Alpha Therapies
Brief Title: A Study to Evaluate the Safety and Efficacy of MabThera (Rituximab) in Combination With Methotrexate (MTX) in Participants With Active Rheumatoid Arthritis Who Failed on Anti-Tumor Necrosis Factor Alpha Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17042; 102-20 (Other: registry identifier)
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (2):
- Placebo Plus Methotrexate (Placebo Comparator): Participants will be administered placebo by intravenous infusion on Days 1 and 15 along with MTX 10-25 mg per os (p.o.) or parenterally once a week up to 24 weeks and will be followed up to Week 104.
  Interventions: Drug: Methotrexate; Other: Placebo
- Rituximab plus Methotrexate (Experimental): Participants will be administered rituximab 1000 mg as intravenous infusion on Days 1 and 15 along with MTX 10-25 mg p.o. or parenterally once a week up to Week 24 and will be followed up to Week 104.
  Interventions: Drug: MabThera/Rituxan; Drug: Methotrexate

INTERVENTIONS:
Drug: MabThera/Rituxan — 1
  Arms: Rituximab plus Methotrexate
Drug: Methotrexate — 2
Other: Placebo — 3
  Arms: Placebo Plus Methotrexate

SUMMARY:
This study will assess the safety and efficacy of rituximab combined with MTX in participants with active rheumatoid arthritis (RA) who have had an inadequate response to anti-Tumor Necrosis (TNF) alpha therapy. The anticipated time in the study is up to 2 years and the target sample size is 500 participants. Eligible participants may receive re-treatment with rituximab under a separate protocol WA17531.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18-80 years of age with active RA for at least 6 months;
* Received treatment for RA on an outpatient basis and experienced an inadequate response or intolerance to treatment with at least 1 anti-TNF alpha therapy (etanercept, infliximab or adalimumab);
* Must have received MTX for a minimum of 12 weeks, with the last 4 weeks, prior to screening at a stable dose;
* Participants with swollen joint count (SJC) and tender joint count (TJC) of at least 8 joints at screening and at randomization;
* Radiographic evidence of at least 1 joint with a definite erosion due to RA;
* Participants of reproductive potential must be using reliable contraceptive methods.

Exclusion Criteria:

* Bone or joint surgery within 8 weeks prior to screening or joint surgery planned within 24 weeks of randomization;
* Class IV functional status of RA;
* Previous treatment within 6 months with intravenous gamma globulin, or the Prosorba column;
* Intraarticular or parenteral corticosteroids within 4 weeks prior to screening visit;
* With a live vaccine within 4 weeks prior to randomization;
* Previous treatment with rituximab or other cell-depleting therapies;
* Concurrent treatment with any disease-modifying anti-rheumatic drug (except for MTX) or any anti-TNF alfa factor or other biologic therapy;
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies;
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders;
* Known contraindications to receiving rituximab;
* Known active bacterial, viral, fungal, mycobacterial or other infection;
* History of recurrent significant infection or history of recurrent bacterial infections;
* Primary or secondary immunodeficiency (history of, or currently active);
* History of cancer, including solid tumors and hematologic malignancies (except basal cell or squamous cell carcinoma of the skin that have been excised and cured);
* Women who are pregnant or breast-feeding;
* History of alcohol, drug or chemical abuse within 6 months prior to screening;
* Neuropathies and neurovasculopathies which might interfere with pain evaluation;
* Participants with poor peripheral venous access;
* Intolerance or contraindications to oral or intravenous corticosteroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2003-05; Primary Completion 2005-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (102):
- United States (57):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fullerton, California
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - Rancho Mirage, California
  - Santa Maria, California
  - Upland, California
  - Danbury, Connecticut
  - Boca Raton, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Orlando, Florida
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Shreverport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Smithtown, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Mayfield, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Amarillo, Texas
  - Dallas, Texas
  - Houston, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Seattle, Washington
  - Spokane, Washington
  - Madison, Wisconsin
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
- France (7):
  - Le Kremlin-Bicêtre
  - Montpellier
  - Paris
  - Rouen
  - Strasbourg
  - Toulouse
  - Tours
- Germany (5):
  - Berlin
  - Dresden
  - Leipzig
  - Ratingen
  - Würzburg
- Ireland (2):
  - Cork
  - Dublin
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (6):
  - Udine, Friuli Venezia Giulia
  - Arenzano, Liguria
  - Genoa, Liguria
  - Brescia, Lombardy
  - Milan, Lombardy
  - Pisa, Tuscany
- Amsterdam, Netherlands
- Norway (4):
  - Drammen
  - Lillehammer
  - Oslo
  - Tromsø
- United Kingdom (6):
  - Cannock
  - Leeds
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Lal P, Su Z, Holweg CT, Silverman GJ, Schwartzman S, Kelman A, Read S, Spaniolo G, Monroe JG, Behrens TW, Townsend MJ. Inflammation and autoantibody markers identify rheumatoid arthritis patients with enhanced clinical benefit following rituximab treatment. Arthritis Rheum. 2011 Dec;63(12):3681-91. doi: 10.1002/art.30596. PMID 22127691
- [Derived] Keystone E, Burmester GR, Furie R, Loveless JE, Emery P, Kremer J, Tak PP, Broder MS, Yu E, Cravets M, Magrini F, Jost F. Improvement in patient-reported outcomes in a rituximab trial in patients with severe rheumatoid arthritis refractory to anti-tumor necrosis factor therapy. Arthritis Rheum. 2008 Jun 15;59(6):785-93. doi: 10.1002/art.23715. PMID 18512710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 520 participants were enrolled in the study conducted from 02 May 2003 and 12 July 2012 in 11 countries.
Pre-assignment Details: Of the total randomized 520 participants who met the eligibility criteria, four did not receive the study treatment and were not included in any analysis population.
Groups:
- Placebo Plus Methotrexate: Eligible participants were administered the placebo by intravenous infusion on Days 1 and 15 along with methotrexate (MTX) 10-25 milligrams (mg) per os (p.o.) or parenterally once a week up to Week 24 and were followed up to Week 104.
- Rituximab Plus Methotrexate: Eligible Participants were administered rituximab 1000 mg as intravenous infusion on Days 1 and 15 along with MTX 10-25 mg p.o. or parenterally once a week up to Week 24 and were followed up to Week 104.
Period: Week 24 Analysis
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Started | 208 | 308
Completed | 111 | 253
Not Completed | 97 | 55
Not completed — Lack of Efficacy | 83 | 37
Not completed — Refused treatment | 5 | 5
Not completed — Adverse Event | 1 | 8
Not completed — Failure to return | 3 | 4
Not completed — Rescue therapy | 2 | 0
Not completed — Incorrect diagnosis and treatment | 0 | 1
Not completed — Due to clinical hold | 1 | 0
Not completed — Went onto rescue therapy | 1 | 0
Not completed — Participant unblinded (clinical hold) | 1 | 0
Period: Week 24 to Week 104 Analysis
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Started | 208 (Participants who completed/not completed Week (W) 24 analysis were entered in W24 to W104 analysis.) | 308 (Participants who completed/not completed W24 analysis were entered in W24 to W104 analysis.)
Completed | 103 | 83
Not Completed | 105 | 225
Not completed — Adverse Event | 2 | 5
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 3 | 12
Not completed — Protocol Violation | 0 | 2
Not completed — Refused treatment | 4 | 7
Not completed — Failure to return | 1 | 2
Not completed — Movement into re-treatment study | 77 | 183
Not completed — Other | 17 | 14

BASELINE CHARACTERISTICS:
Population: Safety population included participants who were randomized and received any part of an infusion of the study drug.
Groups:
- Placebo Plus Methotrexate: Eligible participants were administered placebo by intravenous infusion on Days 1 and 15 along with MTX 10-25 mg p.o. or parenterally once a week up to 24 weeks and were followed up to Week 104.
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate | Total
Number analyzed (Participants) | 208 | 308 | 516
Age, Continuous [Median (Full Range); unit: years] | 55.0 [20 to 79] | 53.0 [20 to 81] | 53.0 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 251 | 419
  Male | 40 | 57 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology 20 Response at Week 24
Description: American College of Rheumatology (ACR) 20 response is defined as >= 20% improvement (reduction) in score compared with baseline for both tender joint count (TJC)-68 joints and swollen joint count (SJC)-66 joints, as well as for 3 of the additional 5 ACR core set variables: Patient's Assessment of Pain over the previous 24 hours using a Visual Analog Scale (VAS) ranging from score 0 (no pain) to 100 (unbearable pain); Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS ranging score 0 (no disease activity) to 100 (maximum disease activity); Health Assessment Questionnaire (HAQ):8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale (0=without any difficulty to 3=unable to do) for a total possible score of 0 (best) to 3 (worst); and acute-phase reactant, either C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Week 24
Population: Intent to treat (ITT) population included all randomized participants who received any part of an infusion of study drug. Participants whom treatment allocation was unblinded and who received treatment prior to randomization were excluded.
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
participants | 36 | 153

2. Secondary Outcome: Number of Participants With an ACR 50 Response at Week 24
Description: ACR 50 response is defined as a >= 50% improvement (reduction) in score compared with baseline for both TJC -68 joints and SJC -66 joints, as well as for 3 of the additional 5 ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a VAS ranging from score '0'=no pain to score '100'=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS ranging from score '0'=no disease activity to score '100'=maximum disease activity; HAQ : Health Assessment Questionnaire (HAQ):which included 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale (0=without any difficulty to 3=unable to do), where the sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst); and acute-phase reactant, either CRP or ESR.
Time Frame: Week 24
Population: The ITT population included all randomized participants who received any part of an infusion of study drug. Participants whom treatment allocation was unblinded and who received treatment prior to randomization were excluded.
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
participants | 11 | 80

3. Secondary Outcome: Number of Participants With ACR 70 Response at Week 24
Description: ACR 70 response is defined as a >= 70% improvement (reduction) in score compared with baseline for both TJC -68 joints and SJC -66 joints, as well as for 3 of the additional 5 ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a VAS ranging from score '0'=no pain to score '100'=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS ranging from score '0'=no disease activity to score '100'=maximum disease activity; HAQ : Health Assessment Questionnaire (HAQ):which included 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale (0=without any difficulty to 3=unable to do), where the sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst); and acute-phase reactant, either CRP or ESR.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
participants | 3 | 37

4. Secondary Outcome: Mean Change From Baseline in Disease Activity Score of 28 Joints at Week 24
Description: The disease activity score (DAS28) is an evaluation index of rheumatoid arthritis. The DAS28 applies a mathematical formula based on the following parameters: 1. TJC-28 joints, 2. SJC -28 joints, 3. ESR or CRP measurement, 4. Participant's judgement on his own overall health (global health [GH]) status expressed by a VAS (0 [no disease activity] to 100 [maximum disease activity]). The mathematical formula is 0.56 × √28TJC + 0.28 × √28SJC + 0.7 x loge ESR + 0.014 × GH. The DAS28 scale ranges from score of 0 to 10, where lower scores indicate best disease control and higher scores indicate worsening of disease. Change from Baseline = difference between the score at Week 24 and the score at Baseline.
Time Frame: From Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
units on a scale | -0.4 (1.17) | -1.9 (1.60)

5. Secondary Outcome: Percentage of Participants With DAS28 Low Disease Activity and DAS28 Remission at Week 24
Description: The DAS28 is an evaluation index of RA. The DAS28 applies a mathematical formula based on the following parameters: 1. TJC- 28 joints, 2. SJC- 28 joints, 3. ESR or CRP measurement, 4. Participant's judgement on his own overall health status (GH) expressed by a visual analogue scale VAS (0 [no disease activity] to 100 [maximum disease activity]). The mathematical formula is 0.56 × √28TJC + 0.28 × √28SJC + 0.7 x loge ESR + 0.014 × GH. The DAS28 scale ranges from score of 0 to 10. A participant was categorized as having low disease activity, if participant's DAS28 score was <= 3.2, and was categorized as having clinical remission if participant's DAS28 score was < 2.6.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
percentage of participants
  Low disease activity | 2 | 15
  Remission | 0 | 9

6. Secondary Outcome: Number of Participants With Good, Moderate, or no European League Against Rheumatism Responses at Week 24
Description: European League Against Rheumatism (EULAR) response is defined based on the DAS28 score and the EULAR response criteria (Van Gestel et al, 1996 and 1999). The DAS28 scale ranges from score of 0 to 10, where lower scores indicate best disease control and higher scores indicate worsening of disease. At a given visit, participants with a DAS28 score of < 3.2 are considered good responders if the change from baseline in their DAS28 score is >1.2. Participants with a DAS28 score >= 3.2 to 5.1 are considered moderate responders if the change from baseline in their DAS28 score is <=1.2 to >=0.6. Participants with DAS28 score >5.1 are considered non-responders if the change from baseline in their DAS28 score is <=1.2 to >=0.6.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
participants
  No response | 157 | 105
  Moderate response | 40 | 149
  Good response | 4 | 44

7. Secondary Outcome: Percentage Change From Baseline in the ACR Core Set (SJC, TJC, Patient's and Physician's Global Assessments, Health Assessment Questionnaire, Pain, C-Reactive Protein, and Erythrocyte Sedimentation Rate) Score
Description: Percentage change in the scores of the following parameters of ACR core set relative to respective baseline scores in both study arms was analyzed : SJC (28 and 66 joints) and TJC (28 and 66 joints), patient's global assessment and physician's global assessment based on disease activity (both are expressed by VAS [0 = no disease activity to 100 = maximum disease activity]), HAQ (based on HAQ disability index [HAQDI]) which included 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale (0=without any difficulty to 3=unable to do), where the sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst), pain assessment using a VAS ranging from score 0 (no pain) to 100 (unbearable pain), CRP concentration, and ESR.
Time Frame: From Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
percent change
  SJC (66) | -5.6 (59.19) | -43.0 (52.65)
  SJC (28) | -7.1 (55.35) | -41.3 (52.77)
  TJC (68) | 7.2 (144.58) | -41.8 (52.39)
  TJC (28) | 15.7 (195.94) | -42.0 (63.47)
  Physician's global assessment | -4.2 (47.23) | -40.8 (39.31)
  Patient's global assessment | -3.1 (44.01) | -25.4 (117.90)
  Patient's pain assessment | 2.8 (55.61) | -23.8 (131.59)
  HAQ | -2.0 (30.46) | -24.3 (34.92)
  CRP | 80.0 (452.94) | -36.3 (80.3)
  ESR | 11.4 (95.95) | -29.3 (59.92)

8. Secondary Outcome: Mean Change From Baseline of Short Form 36 Total Scores at Week 24
Description: The Short Form (SF)-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual daily activities because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems since last month; 7) limitations in usual work (house hold and outside) due to emotional problems 8) current and 1 year past status of health 9) general mental health. Transforming and standardizing these domains leads to the calculation of the physical component summary and mental component summary measures. Scores on each item were summed and averaged (range 0 [worst] to 100 [best]); increase in score from baseline indicated improvement. Change from Baseline = difference between the score at Week 24 and the score at Baseline.
Time Frame: From Baseline (Day 1) to Week 24
Population: The ITT population included all randomized participants who received any part of an infusion of study drug. Participants with available data at the time of evaluation were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 197 | 294
units on a scale
  Physical score | 0.9 (5.65) | 5.8 (8.47)
  Mental health score | 1.3 (9.43) | 4.7 (11.75)

9. Secondary Outcome: Number of Participants With Categorical Change From Baseline in the Physical Component Scores of SF-36
Description: The SF-36 determined participants' overall quality of life by assessing :1) limitations in physical functioning due to health problems; 2) limitations in usual daily activities because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems since last month; 7) limitations in usual work (house hold and outside) due to emotional problems 8) current and 1 year past status of health 9) general mental health. Scores on physical component were summed and averaged (range 0 [worst] to 100 [best]); If participants' had shown change from baseline in physical health component score >5.42, it was considered as improved; score between -5.42 to 5.42 was considered as unchanged, and score < -5.42 was considered as worsened. Change from Baseline = difference between the score of physical component at Week 24 and the score at Baseline.
Time Frame: From Baseline (Day 1) to Week 24
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 197 | 294
participants
  Improved | 25 | 141
  Unchanged | 158 | 136
  Worsened | 14 | 17

10. Secondary Outcome: Number of Participants With Change From Baseline in the Mental Component Scores of SF-36
Description: The SF-36 determined participants' overall quality of life by assessing :1) limitations in physical functioning due to health problems; 2) limitations in usual daily activities because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems since last month; 7) limitations in usual work (house hold and outside) due to emotional problems 8) current and 1 year past status of health 9) general mental health. Scores on mental component were summed and averaged (range = 0 [worst]-100 [best]); increase from baseline indicated improvement. If participants' had shown change from baseline in mental health score >6.33, it was considered as improved; scores between -6.33 to 6.33 was considered unchanged, and score <-6.33 was considered as worsened. Change from Baseline = difference between the mental component score at Week 24 and the score at Baseline.
Time Frame: From Baseline (Day 1) to Week 24
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 197 | 294
participants
  Improved | 40 | 111
  Unchanged | 128 | 144
  Worsened | 29 | 39

11. Secondary Outcome: Mean Change From Baseline in the Genant-modified Sharp Joint Space Narrowing Score, Genant-modified Sharp Total Score, and Erosion Score
Description: The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. Joint space narrowing scores of 0-4 (9 gradations) are assigned to 13 joints in each hand and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140. The maximum joint space narrowing score is 38 x 4.0 = 152. Both the erosion and joint space narrowing scores are normalized to 145 and are added together for a maximum total Genant-modified Sharp score of 290. For all the three radiograph assessment, the minimum score is 0. A higher score indicates more damage and a negative change score indicates improvement. The change in score is to be calculated as: Change from Baseline = difference between the score at Weeks 24, 56, or 104 and the score at Baseline.
Time Frame: From Baseline (Day 1) to Weeks (W) 24, 56, and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 201 | 298
units on a scale
  Sharp-Genant total score, W24, n = 201, 298 | -4.3 (24.09) | -1.2 (20.90)
  Sharp-Genant total score, W56, n = 184, 273 | 2.31 (5.283) | 1.00 (2.751)
  Sharp-Genant total score, W104, n = 186,279 | 2.82 (6.398) | 1.16 (3.429)
  Erosion score, W24, n = 201, 298 | -1.6 (12.15) | -0.4 (10.45)
  Erosion score, W56, n = 184, 273 | 1.32 (3.155) | 0.59 (1.843)
  Erosion score, W104, n = 186,279 | 1.81 (4.187) | 0.73 (2.262)
  Joint space narrowing score, W24, n = 201, 298 | -2.5 (12.71) | -0.9 (10.90)
  Joint space narrowing score, W56, n = 184, 273 | 0.99 (2.571) | 0.41 (1.323)
  Joint space narrowing score, W104, n = 186,279 | 1.01 (2.618) | 0.43 (1.563)

12. Secondary Outcome: Percentage of Participants Without Erosive Progression
Description: The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140 which is normalized to 145. The minimum score is 0 and the maximum score is 145. A higher score indicates more damage and negative change score indicates improvement.
Time Frame: Up to Week 104
Population: ITT population included all randomized participants who received any part of an infusion of study medication. Participants with available data at the time of evaluation were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Number analyzed (Participants) | 187 | 281
percentage of participants
  Baseline to Year 1, n = 186, 278 | 51 | 66
  Year 1 to Year 2, n = 186, 278 | 58 | 73
  Baseline to Year 2, n = 187, 281 | 44 | 60

ADVERSE EVENTS:
Time Frame: Up to Week 104
Description: Adverse events were captured in safety analysis population. Safety population included participants who were randomized and received any part of an infusion of the study drug.
Arm/Group | Placebo Plus Methotrexate | Rituximab Plus Methotrexate
Serious Adverse Events (participants affected / at risk) | 26/208 | 50/308
Other Adverse Events (participants affected / at risk) | 152/208 | 225/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Methotrexate (N=208) | Rituximab Plus Methotrexate (N=308)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Abscess intestinal (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Zoonosis (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 1 | 3
Vasculitis (Vascular disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Synovectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Methotrexate (N=208) | Rituximab Plus Methotrexate (N=308)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 87 | 106
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 16
Upper Respiratory Tract infection (Infections and infestations) | 17 | 36
Nasopharyngitis (Infections and infestations) | 15 | 30
Bronchitis (Infections and infestations) | 15 | 25
Urinary Tract Infection (Infections and infestations) | 15 | 21
Sinusitis (Infections and infestations) | 14 | 12
Headache (Nervous system disorders) | 21 | 31
Dizziness (Nervous system disorders) | 8 | 16
Diarrhoea (Gastrointestinal disorders) | 18 | 21
Nausea (Gastrointestinal disorders) | 8 | 23
Fatigue (General disorders) | 12 | 21
Pyrexia (General disorders) | 7 | 17
Hypertension (Vascular disorders) | 12 | 26
Insomnia (Psychiatric disorders) | 9 | 17
Rash (Skin and subcutaneous tissue disorders) | 9 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights